CLINICAL TRIAL: NCT04821674
Title: A Phase 1/2 Study to Assess the Safety, Immunogenicity and Recommended Dose of DS-5670a (COVID-19 Vaccine) in Japanese Healthy Adults and Elderly Subjects
Brief Title: Study of DS-5670a (COVID-19 Vaccine) in Japanese Healthy Adults and Elderly Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DS5670-A-J101; jRCT2071200110 (Other: Japan Registry of Clinical Trial)
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Covid19
Keywords: COVID-19 Prevention; SARS CoV-2; Coronavirus Vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Cohort A1: DS-5670a 10 µg (Experimental): Healthy adults participants will be randomized to receive a intramuscular injection of DS-5670a 10 µg.
  Interventions: Biological: DS-5670a
- Cohort A2: DS-5670a 30 µg (Experimental): Healthy adults participants will be randomized to receive a intramuscular injection of DS-5670a 30 µg.
  Interventions: Biological: DS-5670a
- Cohort A3: DS-5670a 60 µg (Experimental): Healthy adults participants will be randomized to receive a intramuscular injection of DS-5670a 60 µg.
  Interventions: Biological: DS-5670a
- Cohort A4: DS-5670a 100 µg (Experimental): Healthy adults participants will be randomized to receive a intramuscular injection of DS-5670a 100 µg.
  Interventions: Biological: DS-5670a
- Cohort A: Placebo (Placebo Comparator): Healthy adults participants will be randomized to receive a intramuscular injection of placebo.
  Interventions: Biological: Placebo
- Cohort B1: DS-5670a 10 µg (Experimental): Healthy elderly participants will be randomized to receive a intramuscular injection of DS-5670a 10 µg.
  Interventions: Biological: DS-5670a
- Cohort B2: DS-5670a 30 µg (Experimental): Healthy elderly participants will be randomized to receive a intramuscular injection of DS-5670a 30 µg.
  Interventions: Biological: DS-5670a
- Cohort B3: DS-5670a 60 µg (Experimental): Healthy elderly participants will be randomized to receive a intramuscular injection of DS-5670a 60 µg.
  Interventions: Biological: DS-5670a
- Cohort B4: DS-5670a 100 µg (Experimental): Healthy elderly participants will be randomized to receive a intramuscular injection of DS-5670a 100 µg.
  Interventions: Biological: DS-5670a
- Cohort B: Placebo (Placebo Comparator): Healthy elderly participants will be randomized to receive a intramuscular injection of placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: DS-5670a — DS-5670a (10, 30, 60 or 100 µg) administered as an intramuscular injection into the deltoid muscle of the upper arm; 2 injections total
  Arms: Cohort A1: DS-5670a 10 µg; Cohort A2: DS-5670a 30 µg; Cohort A3: DS-5670a 60 µg; Cohort A4: DS-5670a 100 µg; Cohort B1: DS-5670a 10 µg; Cohort B2: DS-5670a 30 µg; Cohort B3: DS-5670a 60 µg; Cohort B4: DS-5670a 100 µg
Biological: Placebo — Placebo administered as an intramuscular injection into the deltoid muscle of the upper arm; 2 injections total
  Arms: Cohort A: Placebo; Cohort B: Placebo

SUMMARY:
This study will assess the safety, tolerability and immunogenicity of DS-5670a (COVID-19 Vaccine) and determine the recommended dose in Japanese healthy adults and elderly participants.

ELIGIBILITY:
Inclusion Criteria:

* Japanese citizen
* Healthy adults aged ≥20 and <65 years, or healthy elderly aged ≥65 and <75 years (at the time of informed consent)
* Body Mass Index (BMI) is ≥17.5 and <30.0 kg/m^2 (at screening)
* Participants who can follow the compliance requirements during clinical trials, undergo medical examinations and tests specified by the protocol, and report symptoms, etc.

Exclusion Criteria:

* Have a history of immunodeficiency or having a close relative with congenital immunodeficiency.
* Have a history of SARS-CoV-2 infection.
* Have previously participated in an investigational study of SARS-Cov-2 vaccine or involving LNPs.
* Have a history of anaphylaxis or severe allergies due to food, cosmetics, medicines, or vaccination
* Have alcohol or drug dependence.
* Have a fever of ≥39.0°C or symptoms of suspected allergies such as systemic rash within 2 days after past vaccination, etc.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants Reporting Treatment-emergent Adverse Events | Day 1 up to Day 57 post-dose
Number of Participants Reporting Local and Systemic Adverse Events | Day 1 up to Day 14 post-first and second dose
Number of Participants Reporting Serious Events | Day 1 up to 12 months post-second dose
Geometric Mean Titer (GMT) of SARS-CoV-2 Specific Neutralizing Antibody | Days 15, 29, 43, and 57 post-dose
Geometric Mean Fold Rise (GMFR) of SARS-CoV-2 Specific Neutralizing Antibody | Days 15, 29, 43, and 57 post-dose
Seroconversion Rates of SARS-CoV-2 Specific Neutralizing Antibody | Days 15, 29, 43, and 57 post-dose

SECONDARY OUTCOMES:
GMT of anti-IgG Antibody | Days 15, 29, 43, and 57 post-dose
GMFR of anti-IgG Antibody | Days 15, 29, 43, and 57 post-dose
Seroconversion Rates of anti-IgG Antibody | Days 15, 29, 43, and 57 post-dose
Pharmacokinetic Parameter of Maximum (Peak) Observed Plasma Concentration (Cmax) Following Intramuscular Injection of DS-5670a | Days 1, 2, 4, 8, 15, 29, 30, 32, 36, 43, and 57 post-dose
  Cmax of plasma MAFB-7566a and constituent lipids of lipid nanoparticle (LNP) will be assessed.
Pharmacokinetic Parameter of Time to Reach Maximum Concentration (Tmax) Following Intramuscular Injection of DS-5670a | Days 1, 2, 4, 8, 15, 29, 30, 32, 36, 43, and 57 post-dose
  Tmax of plasma MAFB-7566a and constituent lipids of LNP will be assessed.
Pharmacokinetic Parameter of Area Under the Concentration-time Curve Following Intramuscular Injection of DS-5670a | Days 1, 2, 4, 8, 15, 29, 30, 32, 36, 43, and 57 post-dose
  Area under the concentration-time curve from time 0 to last measurable time point (AUClast) and time 0 to infinity (AUCinf) of plasma MAFB-7566a and constituent lipids of LNP will be assessed.
Pharmacokinetic Parameter of Apparent Total Body Clearance (CL/F) Following Intramuscular Injection of DS-5670a | Days 1, 2, 4, 8, 15, 29, 30, 32, 36, 43, and 57 post-dose
  CL/F of plasma MAFB-7566a and constituent lipids of LNP will be assessed.
Pharmacokinetic Parameter of Terminal Elimination Half-life (t1/2) Following Intramuscular Injection of DS-5670a | Days 1, 2, 4, 8, 15, 29, 30, 32, 36, 43, and 57 post-dose
  Half-life (t1/2) of plasma MAFB-7566a and constituent lipids of LNP will be assessed.
Pharmacokinetic Parameter of Apparent Volume of Distribution (Vz/F) Following Intramuscular Injection of DS-5670a | Days 1, 2, 4, 8, 15, 29, 30, 32, 36, 43, and 57 post-dose
  Vz/F of plasma MAFB-7566a and constituent lipids of LNP will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (1):
- SOUSEIKAI Hakata Clinic, Hakata, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No